CLINICAL TRIAL: NCT02686073
Title: Revising the Norms of Labor Progress in Egyptian Nulliparous Women in Relation to Maternal Body Mass Index Categories
Brief Title: Effect of Maternal Body Mass Index on Labor Progress in Nulliparous Women
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Shafie Belal, Lecturer, Cairo University
Other Study IDs: Kasr El-Aini Hospital
Record Dates: First submitted 2016-02-07; First posted 2016-02-19 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Labor Progress
Keywords: BMI; progress of labor; nulliparous women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group A: Underweight participants whose body mass index is less than 18.5 kg/m2
- Group B: Control group, in which the participants belong to the normal body mass index range , from 18.5 to 29.9 kg/m2
- Group C: Obese participants whose body mass index is more than or equal to 30 kg/m2.

SUMMARY:
Study the rate of progress of labor among nulliparous women belonging to different body mass index groups, & observe how does this variation in maternal body mass index may affect the course of labor.

DETAILED DESCRIPTION:
For nulliparous cases presenting to the labor ward, maternal height & weight will be collected at the time of admission to calculate the BMI (body mass index) & further classified according to WHO (World Health Organization) categories. Putting into consideration the physiological increase in BMI related to pregnancy, the overweight participants whose BMI (25-29.9) will be combined with the normal range BMI (18.5-24.9) category. Labor characteristics of these participants will be then compared with those of the underweight (BMI less than 18.5) & obese (BMI 30 or higher) participants.Females are assigned in one of 3 groups based on their BMI; Underweight group (BMI <18.5kg/m2), Control group whose BMI within normal range (18.5-29.9 kg/m2),& Obese group (BMI more than or equal 30kg/m2).

Labor management protocols are fixed. Data on labor progression are collected, including cervical dilatation, cervical effacement, head station & descent. The median duration of labor , estimated by rate of cervical dilatation in cm, will be used as a measurement of labor progression in each group.

A cesarean section for abnormal labor pattern will be documented as failure of progress.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women in active phase of labor, with an age range from 20 to 40 years.

Full term pregnancy, singleton, viable fetus, cephalic (vertex) presentation, occipito-anterior position.

Exclusion Criteria:

* Multiparous women. Preterm labor. Passed date delivery. Multiple gestation. Large fetal weight (more than 4000g). Intrauterine fetal death. Intrauterine fetal growth restriction. Major fetal congenital anomalies. Rupture of membranes before onset of active labor. Fetal malposition or malpresentation. Inadequate pelvis or cephalopelvic disproportion. Maternal medical disorder.

Induction of labor by oxytocin or prostaglandins. Conditions requiring urgent delivery eg antepartum haemorrhage, fetal distress, cord prolapse.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant nulliparous women, at term, during labor
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-02-20 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
rate of cervical dilatation | every 2 hours during active phase of labor, from admission to the labor ward until second stage of labor.
  in centimeters

SECONDARY OUTCOMES:
descent of fetal head | every 2 hours during active phase of labor, from admission to the labor ward until second stage of labor
  head station

OTHER OUTCOMES:
duration of active phase of labor | all through the course of labor, individually assessed for each participant, starting from the time of admission to labor ward until start of second stage of labor
  total duration in hours
duration of second stage of labor | from start of second stage of labor ( full cervical dilatation) until delivery of fetus
  total duration in minutes
mode of delivery | labor
  vaginal delivery or cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Sh Belal, hospital, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Belal DS, Marie HM, Rashwan H, Abdelaziz S, Gabr AA, Elzayat AR. Prospective study of the effect of maternal body mass index on labor progress in nulliparous women in Egypt. Int J Gynaecol Obstet. 2017 Dec;139(3):329-335. doi: 10.1002/ijgo.12322. Epub 2017 Oct 3. PMID 28886213